CLINICAL TRIAL: NCT01461187
Title: Effects in Type of Birth of Physical Exercise During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Servidor Publico Estadual (Other)
Collaborators: Maternal Breastfeeding Incentive Center (CIAMA) (Unknown)
Responsible Party: Principal Investigator, Lilian Cristina da Silveira, Physiotherapist master's degree in health sciences, Hospital do Servidor Publico Estadual
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Líliancsilveira
Record Dates: First submitted 2011-10-04; First posted 2011-10-27 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Pregnancy
Keywords: Exercise; Pregnancy; Childbirth; Vaginal; Cesarean section
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- exercise in pregnancy (Experimental): 37 pregnant women who performed supervised aerobic physical exercises twice a week
  Interventions: Other: exercise during pregnancy
- Control group (No Intervention): 29 pregnant women who had not performed any kind of physical activity during pregnancy

INTERVENTIONS:
Other: exercise during pregnancy — supervised aerobic physical exercises twice a week.
  Arms: exercise in pregnancy

SUMMARY:
Abstract:

Objectives:[The goal is] to confirm if physical activity of medium intensity performed during gestation can influence the way of delivery, and observe the adherence to exercise among pregnant women with different education levels. Methods: Held at the Center for Breastfeeding Incentive in the city of São Sebastião, State of São Paulo (Brazil), between April 7, 2008 and April 14, 2009, the prospective study involved 66 primigravid women, who were divided into two groups: the exercise group (GE) that exercised regularly during pregnancy, and the other control group (GC) that did not exercise regularly during same period. The significance level adopted in this study was five per cent (p = 0.05).

DETAILED DESCRIPTION:
Research was conducted at the Maternal Breastfeeding Incentive Center (Centro de Incentivo ao Aleitamento Materno - CIAMA) in São Sebastião, São Paulo, Brazil. The 66 primigravidas were allocated to two groups: a control group, with 29 pregnant women who had not performed any kind of physical activity during pregnancy, and another group, the exercise group, with 37 pregnant women who performed supervised aerobic physical exercises twice a week. These volunteers needed to attend at least 20 sessions to be included in the research. No pregnant women in the control group or the exercise group had performed regular physical activity in the year prior to the pregnancy. All participants received verbal information on how the research would be conducted, and after agreeing to participate they signed a free and informed consent term. The physical activity was prescribed by a physical therapist who remained available to address any doubts about the physical activity and about the research. The study followed the baselines of the American Congress of Obstetricians and Gynecologists (ACOG), where the environment temperature hasn't exceeded 28 °C. The pregnant women were told to wear comfortable clothes and to drink water before and during the activity, and not to perform physical activity while fasting. They were also instructed to interrupt the activity in case they felt dizziness, breathlessness, pain, muscle weakness, dyspnea prior to effort or in case they presented calf swelling or pain, bleeding or signs of labor, or, still, if they noticed decrease in fetal movements. Two weeks after birth the volunteers were contacted by phone to collect information on the type of birth.

ELIGIBILITY:
The inclusion criteria:

* nulliparae,
* sedentary women,
* ages between 18 and 30,
* gestation age superior to 18 weeks without clinical or obstetrical complications

Exclusion Criteria:

The volunteers in the GE couldn't have a gestation age superior to 20 weeks, had to participate on regular physical activity twice a week, and have a total frequency of at least 20 sessions. The EG pregnant women with frequency inferior to 20 sessions were discarded from the study.

The volunteers in the CG couldn't have performed regular physical activity during pregnancy. In both groups, the participants hadn't performed regular physical activity in the year prior to the pregnancy.

However, 31 women were discarded during the research: three for miscarriage, being two from the GE and one from the GC; one from the GE for anemia; one from the GC for pre-eclampsia; two for loss of contact after birth, being one from each group; 11 from the GE for not reaching the minimum frequency; seven claimed personal reasons for leaving the research, being five from the GC and two from the GE; and six participants abandoned the study.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Predomination of type of birth, vaginal birth or Cesarean section among pregnant women participating in the exercise group and the control group. | Research conducted between April 7, 2008 and April 14, 2009 (one year)
  Of the 66 volunteers, 37 were part of the exercise group (EG) and 29 of the control group (CG). Of the 37 in the control group, 25 had vaginal birth, while 12 had a Cesarean. In contrast, of the 29 in the CG, 11 had vaginal birth and 18 had a Cesarean.

SECONDARY OUTCOMES:
Adhesion to exercise among the pregnant women with undergraduate and elementary education. | The investigation lasted for one year
  Of the 66 volunteers, 12 had undergraduate education. Of these, 11 were part of the EG and one of the CG. In contrast, 15 of the 66 pregnant volunteers had primary education, six of which were part of the EG, while nine were part of the CG.

CONTACTS AND LOCATIONS:
Overall Officials: Lílian Cristina da Silveira, Principal Investigator — hostital public servant's state sao paulo (HSPE)
Locations (1):
- center of encouraging breastfeeding (CIAMA), São Sebastião, São Paulo, Brazil

REFERENCES:
- [Background] Villar J, Carroli G, Zavaleta N, Donner A, Wojdyla D, Faundes A, Velazco A, Bataglia V, Langer A, Narvaez A, Valladares E, Shah A, Campodonico L, Romero M, Reynoso S, de Padua KS, Giordano D, Kublickas M, Acosta A; World Health Organization 2005 Global Survey on Maternal and Perinatal Health Research Group. Maternal and neonatal individual risks and benefits associated with caesarean delivery: multicentre prospective study. BMJ. 2007 Nov 17;335(7628):1025. doi: 10.1136/bmj.39363.706956.55. Epub 2007 Oct 30. PMID 17977819
- [Background] Gerten KA, Coonrod DV, Bay RC, Chambliss LR. Cesarean delivery and respiratory distress syndrome: does labor make a difference? Am J Obstet Gynecol. 2005 Sep;193(3 Pt 2):1061-4. doi: 10.1016/j.ajog.2005.05.038. PMID 16157112
- [Background] Chalmers B. WHO appropriate technology for birth revisited. Br J Obstet Gynaecol. 1992 Sep;99(9):709-10. doi: 10.1111/j.1471-0528.1992.tb13867.x. PMID 1420006
- [Background] Bungum TJ, Peaslee DL, Jackson AW, Perez MA. Exercise during pregnancy and type of delivery in nulliparae. J Obstet Gynecol Neonatal Nurs. 2000 May-Jun;29(3):258-64. doi: 10.1111/j.1552-6909.2000.tb02047.x. PMID 10839574
- [Background] Cavalcante SR, Cecatti JG, Pereira RI, Baciuk EP, Bernardo AL, Silveira C. Water aerobics II: maternal body composition and perinatal outcomes after a program for low risk pregnant women. Reprod Health. 2009 Jan 6;6:1. doi: 10.1186/1742-4755-6-1. PMID 19126239
- [Background] Zeanah M, Schlosser SP. Adherence to ACOG guidelines on exercise during pregnancy: effect on pregnancy outcome. J Obstet Gynecol Neonatal Nurs. 1993 Jul-Aug;22(4):329-35. doi: 10.1111/j.1552-6909.1993.tb01813.x. PMID 8410432
- [Background] ACOG Committee Obstetric Practice. ACOG Committee opinion. Number 267, January 2002: exercise during pregnancy and the postpartum period. Obstet Gynecol. 2002 Jan;99(1):171-3. doi: 10.1016/s0029-7844(01)01749-5. PMID 11777528
- [Background] Artal R, O'Toole M. Guidelines of the American College of Obstetricians and Gynecologists for exercise during pregnancy and the postpartum period. Br J Sports Med. 2003 Feb;37(1):6-12; discussion 12. doi: 10.1136/bjsm.37.1.6. No abstract available. PMID 12547738
- [Background] Juhl M, Andersen PK, Olsen J, Madsen M, Jorgensen T, Nohr EA, Andersen AM. Physical exercise during pregnancy and the risk of preterm birth: a study within the Danish National Birth Cohort. Am J Epidemiol. 2008 Apr 1;167(7):859-66. doi: 10.1093/aje/kwm364. Epub 2008 Feb 25. PMID 18303008
- [Background] San Juan Dertkigil M, Cecatti JG, Sarno MA, Cavalcante SR, Marussi EF. Variation in the amniotic fluid index following moderate physical activity in water during pregnancy. Acta Obstet Gynecol Scand. 2007;86(5):547-52. doi: 10.1080/00016340601181649. PMID 17464582
- [Background] Liu J, Laditka JN, Mayer-Davis EJ, Pate RR. Does physical activity during pregnancy reduce the risk of gestational diabetes among previously inactive women? Birth. 2008 Sep;35(3):188-95. doi: 10.1111/j.1523-536X.2008.00239.x. PMID 18844644
- [Background] Kardel KR, Kase T. Training in pregnant women: effects on fetal development and birth. Am J Obstet Gynecol. 1998 Feb;178(2):280-6. doi: 10.1016/s0002-9378(98)80013-6. PMID 9500487
- [Background] Santos IA, Stein R, Fuchs SC, Duncan BB, Ribeiro JP, Kroeff LR, Carballo MT, Schmidt MI. Aerobic exercise and submaximal functional capacity in overweight pregnant women: a randomized trial. Obstet Gynecol. 2005 Aug;106(2):243-9. doi: 10.1097/01.AOG.0000171113.36624.86. PMID 16055571
- [Background] Garshasbi A, Faghih Zadeh S. The effect of exercise on the intensity of low back pain in pregnant women. Int J Gynaecol Obstet. 2005 Mar;88(3):271-5. doi: 10.1016/j.ijgo.2004.12.001. Epub 2005 Jan 16. PMID 15733880
- [Background] Morkved S, Bo K, Schei B, Salvesen KA. Pelvic floor muscle training during pregnancy to prevent urinary incontinence: a single-blind randomized controlled trial. Obstet Gynecol. 2003 Feb;101(2):313-9. doi: 10.1016/s0029-7844(02)02711-4. PMID 12576255
- [Background] Exercise during pregnancy and the postpartum period. ACOG Technical Bulletin Number 189--February 1994. Int J Gynaecol Obstet. 1994 Apr;45(1):65-70. PMID 7913067
- [Background] Watson WJ, Katz VL, Hackney AC, Gall MM, McMurray RG. Fetal responses to maximal swimming and cycling exercise during pregnancy. Obstet Gynecol. 1991 Mar;77(3):382-6. PMID 1992404
- [Background] Dwarkanath P, Muthayya S, Vaz M, Thomas T, Mhaskar A, Mhaskar R, Thomas A, Bhat S, Kurpad A. The relationship between maternal physical activity during pregnancy and birth weight. Asia Pac J Clin Nutr. 2007;16(4):704-10. PMID 18042532
- [Background] Ellington C, Katz VL, Watson WJ, Spielman FJ. The effect of lateral tilt on maternal and fetal hemodynamic variables. Obstet Gynecol. 1991 Feb;77(2):201-3. doi: 10.1097/00006250-199102000-00007. PMID 1988881
- [Background] Salles-Costa R, Werneck GL, Lopes CS, Faerstein E. [The association between socio-demographic factors and leisure-time physical activity in the Pro-Saude Study]. Cad Saude Publica. 2003 Jul-Aug;19(4):1095-105. doi: 10.1590/s0102-311x2003000400031. Epub 2003 Sep 8. Portuguese. PMID 12973574
- [Background] Fell DB, Joseph KS, Armson BA, Dodds L. The impact of pregnancy on physical activity level. Matern Child Health J. 2009 Sep;13(5):597-603. doi: 10.1007/s10995-008-0404-7. Epub 2008 Aug 22. PMID 18719984
- [Result] Shearer EL. Cesarean section: medical benefits and costs. Soc Sci Med. 1993 Nov;37(10):1223-31. doi: 10.1016/0277-9536(93)90334-z. PMID 8272901
- See also: link related to support groups for normal delivery — http://www.partodoprincipio.com.br